CLINICAL TRIAL: NCT04759807
Title: A Phase 1b 3-way Crossover Study to Assess the Safety, Tolerability and Pharmacokinetics of Repeated Once Daily Doses of PUR1800 in Adult Patients With Stable Chronic Obstructive Pulmonary Disease
Brief Title: A Phase 1b Study of PUR1800 in Patients With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 601-0016
Record Dates: First submitted 2021-02-01; First posted 2021-02-18 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: PUR1800, or placebo is dosed daily for 14 consecutive days in adult subjects with stable COPD over three discrete TPs. Subjects will be randomised to one of the following 3 treatment sequences: Sequence Period 1 Period 2 Period 3
  1. Placebo PUR1800 250 μg PUR1800 500 μg
  2. PUR1800 250 μg Placebo PUR1800 500 μg
  3. PUR1800 250 μg PUR1800 500 μg Placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: A computerised randomisation scheme will be created and shall be considered blinded. The randomisation is available only to the clinical research unit pharmacy staff that are preparing the drug who will not be involved in any other aspect of the study including administration of the drug. It will not be made available to the subjects, site(s) PI(s), or members of the staff responsible for the monitoring and evaluation of safety assessments. PUR1800 and placebo capsules will be of the same shape, size, and color to ensure that the blind is maintained. A subject's treatment assignment will only be unblinded when knowledge of the treatment is essential for the further clinical management of the subject on this study or may potentially impact the safety of subjects currently enrolled or subjects in subsequent enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo designed for administration in the proposed clinical study consists of a dry powder composed of the same excipients as the active (sodium sulfate, mannitol and polysorbate 80), pre-metered into HPMC capsules at the same 5 mg powder fill weight as the active formulations. Subjects will receive 14 doses administered once daily in the morning.
  Interventions: Drug: Placebo Comparator
- PUR1800 250 μg (Active Comparator): The PUR1800 drug product intended for use in the proposed clinical study comprises bulk powder containing 5 wt% or 10 wt% RV1162 pre-metered into HPMC capsules for oral delivery via a passive DPI. The capsules contain 5 milligrams (mg) of the powder formulation, corresponding to 250 μg and 500 μg nominal dose strengths of RV1162. Subjects will receive 14 doses administered once daily in the morning.
  Interventions: Drug: PUR1800 250 ug
- PUR1800 500 μg (Active Comparator): The PUR1800 drug product intended for use in the proposed clinical study comprises bulk powder containing 5 wt% or 10 wt% RV1162 pre-metered into HPMC capsules for oral delivery via a passive DPI. The capsules contain 5 milligrams (mg) of the powder formulation, corresponding to 250 μg and 500 μg nominal dose strengths of RV1162. Subjects will receive 14 doses administered once daily in the morning.
  Interventions: Drug: PUR1800 500 ug

INTERVENTIONS:
Drug: Placebo Comparator — The placebo designed for administration in the proposed clinical study consists of a dry powder composed of the same excipients as the active (sodium sulfate, mannitol and polysorbate 80), pre-metered into HPMC capsules at the same 5 mg powder fill weight as the active formulations. Subjects will receive 14 doses administered once daily in the morning.
  Arms: Placebo
Drug: PUR1800 250 ug — The PUR1800 drug product intended for use in the proposed clinical study comprises bulk powder containing 5 wt% or 10 wt% RV1162 pre-metered into HPMC capsules for oral delivery via a passive DPI. The capsules contain 5 milligrams (mg) of the powder formulation, corresponding to a 250 μg nominal dose strength of RV1162. Subjects will receive 14 doses administered once daily in the morning.
  Arms: PUR1800 250 μg
Drug: PUR1800 500 ug — The PUR1800 drug product intended for use in the proposed clinical study comprises bulk powder containing 5 wt% or 10 wt% RV1162 pre-metered into HPMC capsules for oral delivery via a passive DPI. The capsules contain 5 milligrams (mg) of the powder formulation, corresponding to a 500 μg nominal dose strength of RV1162. Subjects will receive 14 doses administered once daily in the morning.
  Arms: PUR1800 500 μg

SUMMARY:
This is a randomised, placebo-controlled, double-blind 3-way crossover study in which PUR1800, or placebo is dosed daily for 14 consecutive days in adult subjects with stable COPD over three discrete TPs. Subjects will be randomised to one of the following 3 treatment sequences:

Sequence Period 1 Period 2 Period 3

1. Placebo PUR1800 250 μg PUR1800 500 μg
2. PUR1800 250 μg Placebo PUR1800 500 μg
3. PUR1800 250 μg PUR1800 500 μg Placebo

Since this is the first study in humans in which the iSPERSE formulation is being administered, the 3 treatment sequences are designed in order to ensure that the lower dose of PUR1800 (250 μg) is administered prior to the administration of the higher dose of PUR1800 (500 μg).

DETAILED DESCRIPTION:
The study design is as follows

Informed Consent: Before any study specific procedures are conducted or study requirements are expected of a patient, the patient must review and sign an IEC-approved informed consent form.

Screening: Subjects will be screened for eligibility to participate in the study within 28 days before randomisation (i.e. TP1, Day 1).

Treatment Periods:

Period 1: On Day 1 all subjects who are eligible for entry into the study will be randomised to 1 of 3 treatment sequences and receive either placebo or the lowest nominal dose of PUR1800 (PUR1800 250 μg) for 14 consecutive days.

Period 2: Following a washout period of at least 28 days after the completion of Period 1 dosing, subjects will receive a treatment other than what the subject received during Period 1 for 14 consecutive days.

Period 3: Following a washout period of at least 28 days after the completion of Period 2 dosing, subjects will receive the treatment that the subject had not received during Periods 1 or 2 (either placebo or PUR1800, 500 μg) for 14 consecutive days.

End of Study (EOS): Subjects will return to the study site 28 days after the last dose of the last TP (or in the event of early withdrawal after the last dose received, if possible) for an EOS visit. Unscheduled visits are permitted at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following:

1. Male or female patients aged 40 to 75 years of age with a body mass index

   ≥ 17 and ≤ 35 kg/m2.
2. Female patients must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method (See Section 9.4.1).
3. Male patients with female partners of childbearing potential must be vasectomised with documented medical assessment of the surgical success or use highly effective contraception together with their female partner(s) (See Section 9.4.1).
4. Female patients must agree not to donate ova/oocytes during the study and for 30 days after the last dose of IMP.
5. Male patients must agree not to donate semen during the study and for 90 days after the last dose of IMP.
6. Confirmed diagnosis by a physician of COPD with symptoms compatible with COPD for at least 1 year prior to screening.
7. Severity of Disease: patients who conform to the current severity classification for GOLD Grade II/III disease in terms of post-bronchodilator spirometry at screening: Post-salbutamol FEV1/FVC ratio of < 0.70. Post-salbutamol FEV1 ≥ 40 % and ≤ 80 % of predicted normal values (based on the Global Lung Function Initiative [GLI-2012][1]).
8. Current or previous tobacco smoker with a smoking history of ≥ 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent).
9. Vital signs recorded from automated blood pressure equipment within the following normal ranges: Blood pressure; systolic value of 90 mmHg to 160 mmHg, diastolic value of 60 mmHg to 90 mmHg and pulse rate ≥ 60 and

   ≤100 beats per minute at screening and prior to randomisation.
10. Able to provide written Informed Consent Form (ICF) prior to participation in any study-related activities, and to comply with the requirements of the study.
11. Able to perform technically acceptable spirometry at screening.
12. Able to produce a sputum sample of adequate quality at either the Screening or Baseline visit prior to randomisation.
13. Able to demonstrate the correct inhalation technique for use of the delivery device and to generate sufficient peak inspiratory flow (PIF) (at least 40 L/min) using the In-Check DIAL device at screening and prior to randomisation.

Exclusion Criteria:

Patients who meet any of the following are not eligible:

1. Upper or lower respiratory tract infection within 6 weeks prior to screening or prior to randomisation.
2. COPD exacerbation requiring oral steroids and/or antibiotics, within the 6 weeks prior to screening or prior to randomisation.
3. Clinically significant abnormal laboratory values at screening that, in the opinion of the investigator would make the patient inappropriate for the study or put the patient at undue risk, specifically liver function tests (LFTs: aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma-glutamyl transferase [GGT], total bilirubin) >3 x upper limit of normal (ULN); hemoglobin <10 gm/dL; absolute neutrophil count (ANC) <1000; white blood cells (WBC) >20,000; Platelets <100,000 and >500,000; prothrombin time (PT) >14 seconds.
4. QTcF of >450 msec in males or >470 msec in females on any of the three individual ECG measurements at screening or prior to randomisation.
5. History of drug or alcohol abuse within the past 2 years prior to screening or prior to randomisation.
6. History of regular alcohol consumption within 6 months prior to screening or prior to randomisation defined as an average weekly intake of >21 units for males, or >14 units for females, where one unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
7. Positive alcohol breath test result at screening or prior to randomisation.
8. Positive urine drugs of abuse test result (unless in the opinion of the investigator this can be explained by the patient's current medications) at screening or prior to randomisation; unexpected or unexplained positive results may require discussion with Sponsor.
9. Current users of e-cigarettes and those who have used these products within one month prior to screening or between screening and randomisation.
10. Known sensitivity to the study drug or any of the excipients of the formulation, or history of clinically significant sensitivity to any agent that, in the opinion of the investigator, would make participation in the study inadvisable.
11. Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug, or intention to donate blood or blood products during the study.
12. Participated in an interventional study involving an experimental therapeutic agent within 3 months of screening or prior to randomisation.
13. Women who have a positive serum β-human chorionic gonadotropin (hCG) pregnancy test at screening or a positive urinary hCG pregnancy test prior to randomisation, is pregnant, lactating, or planning to become pregnant during the study.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or HIV results. Patients who are HBs antibody positive or HB core antibody positive are not excluded provided the HBsAg result is negative. Patients who are HCV Ab positive are not excluded if a subsequent HCV RNA test is negative.
15. Planned surgery or procedures during the participation of the study and for 28 days after the conclusion of study participation.
16. Employee of the investigator or study centre with direct involvement in the proposed study or other studies under the direction of that investigator or study centre, as well as family members of the employees or the investigator.
17. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
18. The patient is unable or unwilling to comply fully with the study protocol.
19. Patient is mentally or legally incapacitated.
20. Unable or unwilling to undergo multiple venepuncture procedures or the patient has poor access to veins suitable for cannulation.
21. Any other reason that, in the opinion of the investigator, would make participation in the study inadvisable.
22. A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation within the last 5 years.
23. A history of > 1 hospitalisation for COPD in the previous 1 year prior to screening.
24. Evidence of cor pulmonale or clinically significant pulmonary hypertension.
25. Requires routine treatment for COPD using one (or more) of the following therapies within the 6 weeks before screening or prior to randomisation: Oral Beta-2 agonists Methyl xanthines Phosphodiesterase (PDE) inhibitors Oral leukotriene inhibitors Oral or parenteral glucocorticoids Antibiotic therapies for acute infections (Note: chronic antibiotic use for prophylaxis, e.g. macrolides, is acceptable).
26. Other respiratory disorders: Patients with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, known alpha-1 antitrypsin deficiency or other active pulmonary diseases other than COPD.
27. Patients with a history of chronic uncontrolled disease including, but not limited to, cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, hematologic, urologic, immunologic, or ophthalmic diseases that, in the opinion of the investigator, would make participation in the study inadvisable.
28. Patients with a history of sleep apnoea requiring non-invasive ventilation or supplemental oxygen during sleep.
29. Previous lung resection or lung reduction surgery.
30. Active participation in a pulmonary rehabilitation program.
31. Has had major surgery within 6 weeks prior to screening or prior to randomisation.
32. A disclosed history, or one known to the Investigator, of significant noncompliance in previous investigational studies or with prescribed medications.
33. History of unstable or uncontrolled hypertension or has been diagnosed with hypertension in last 3 months prior to screening or prior to randomisation.
34. Requires supplemental oxygen, even on an occasional basis.
35. Received a live vaccine within 6 weeks prior to screening or prior to randomisation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events adult patients with stable COPD. | Day 1 through Day 28
  Review of adverse events
Incidence of intraday FEV1 declines (from pre-dose to post-dose) of ≥10%, ≥15%, and ≥20% adult patients with stable COPD. | Day 1 through Day 28
  Review of spirometry data
Respiratory rate | Day 1 through Day 28
  Breaths per minute
Blood presuure | Day 1 through Day 28
  Systolic pressure over diastolic pressure
Heart rate | Day 1 through Day 28
  Beats per minute
Oxygen saturation | Day 1 through Day 28
  As a percentage
Medical history findings | Day 1 through Day 28
  Medical record review
Physical examination findings | Day 1 through Day 28
  Physician's notes
Clinical laboratory parameters | Day 1 through Day 28
  Lab reports with any out of range results flagged
12-Lead ECG findings | Day 1 through Day 28
  ECG report and tracing
Occurrence of PEFR decline of ≥ 30% from the established baseline PEFR | Day 1 through Day 28
  Review of spirometry data
Occurrence of administration of more than 12 inhalations of salbutamol per day over two consecutive days | Day 1 through Day 28
  Review of concomitant medications administered

SECONDARY OUTCOMES:
AUC0-t | Day 1 through Day 14
  Derived from plasma PK samples taken
AUCinf inhaled PUR1800 in adult patients with stable COPD. | Day 1 through Day 14
  Derived from plasma PK samples taken
CL | Day 1 through Day 14
  Derived from plasma PK samples taken
Vss | Day 1 through Day 14
  Derived from plasma PK samples taken
t1/2 | Day 1 through Day 14
  Derived from plasma PK samples taken
Cmax | Day 1 through Day 14
  Derived from plasma PK samples taken
tmax | Day 1 through Day 14
  Derived from plasma PK samples taken
Accumulation factor | Day 1 through Day 14
  Derived from plasma PK samples taken

OTHER OUTCOMES:
Sputum RV1162 concentration | at trough on Days 2, 7, 14, and at the baseline visits prior to TP2 and TP3 as well as the EOS visit after TP3.
  From sputum samples obtained from subject through sputum induction

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Prof, Principal Investigator — The Medicines Evaluation Unit
Locations (1):
- Medicines Evaluation Unit Ltd., Manchester, Wythenshawe, United Kingdom